CLINICAL TRIAL: NCT02822833
Title: The Role of Indocyanine Green to Identify Sentinel Lymph Node in Uterine Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, salih taskin, Assoc. Prof., Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04
Record Dates: First submitted 2016-06-24; First posted 2016-07-04 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Endometrial Neoplasm
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sentinel lymph node mapping (Experimental): Sentinel lymph node mapping with indocyanine green injection to cervix in endometrial cancer patients operated laparoscopically
  Interventions: Procedure: Sentinel lymph node mapping

INTERVENTIONS:
Procedure: Sentinel lymph node mapping — Before laparoscopic hysterectomy and lymphadenectomy procedure for endometrial cancer, Indocyanine green solution will be injected through cervix. Then the surgeon will look for sentinel lymph nodes under fluorescence visualization.
  Other Names: Karl Storz ICG system, to visualize the fluorescence; Indocyanine green, PULSION medical systems

SUMMARY:
Endometrial cancer is the most common gynecologic malignancy in developed countries and the second one in developing countries following cervical cancer. The primary treatment for endometrial cancer involves total hysterectomy and bilateral salpingo-oophorectomy, with adjuvant radiotherapy and/or chemotherapy reserved for patients with advanced disease or who have risk factors for relapse. The tumor is confined to the uterus in 85% of endometrial cancers. Hence, it's controversial to perform systematic lymphadenectomy to all patients. The primary purpose of the present study is the to investigate the feasibility of sentinel lymph node determination in endometrial cancer patients operated via conventional laparoscopy. To determine sentinel lymph nodes cervical indocyanine green will be injected prior to the surgery. During the surgery using fluorescent imaging systems sentinel lymph nodes will be removed and examined by frozen section. Afterwards, systematic pelvic lymphadenectomy will be performed. In case of type II endometrial cancer, grade 3, metastatic sentinel lymph nodes or macroscopically enlarged paraaortic lymph nodes, paraaortic lymphadenectomy will also be performed. The secondary purpose of the study is to compare the conventional laparoscopy in sentinel lymph node mapping of endometrial cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of endometrial cancer
* Clinical stage I or II

Exclusion Criteria:

* Contraindications for operation (hematological or coagulation disorders)
* Advanced stage
* Pregnancy or puerperium
* Fertility preserving surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of sentinel lymph node frozen section | 6 months
Unilateral or bilateral sentinel lymph node detection rate by indocyanine green | 6 months

SECONDARY OUTCOMES:
Negative and positive predictive values for sentinel lymph node frozen section | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School of Medicine Department of Ob&Gyn, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided